CLINICAL TRIAL: NCT05181241
Title: An Open-label Study of Pharmacokinetics, Safety and Tolerability of Drug DD217, Enteric-coated Tablets, 10 mg, Developed by PharmaDiall Ltd (Moscow), on Healthy Volunteers Receiving Single Dose in Fasting State (Phase I)
Brief Title: A Study of Pharmacokinetics, Safety and Tolerability of Dimolegin (DD217)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaDiall Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KI-01-2016
Record Dates: First submitted 2021-12-03; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteers
Keywords: Dimolegin; Dioxaban; DD217; Factor Xa Inhibitor; anticoagulant; therapeutic anticoagulation; thromboprophylaxis; anticoagulation; healthy
MeSH Terms: interventions — (+-)-(1'R*,2'S*,6'R*)-(2-hydroxy-4,6-dimethoxyphenyl)(3'-methyl-2'-(3''-methylbut-2''-enyl)-6-phenylcyclohex-3'-enyl)methanone

STUDY DESIGN:
Intervention Model Description: The study is single center, open-label, prospective, non-randomized with sequential enrollment of volunteers with dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group No. 1 (n=6) Dimolegin - 20 mg (Experimental): Group No. 1 (n=6) consisted of 2 cohorts with 3 volunteers per each. Volunteers of Cohorts 1 and 2 received Dimolegin (DD217) once at a dose of 20 mg
  Interventions: Drug: Dimolegin
- Group No. 2 (n=6) Dimolegin - 40 mg (Experimental): Group No. 2 (n=6) consisted of 2 cohorts with 3 volunteers per each. Volunteers of Cohorts 3 and 4 received Dimolegin (DD217) once at a dose of 40 mg
  Interventions: Drug: Dimolegin
- Group No. 3 (n=12) Dimolegin - 60 mg (Experimental): Group No. 3 (n=12) consisted of 3 cohorts. Cohorts 5 and 6 included 3 volunteers per each, and Cohort 7 included 6 volunteers. All Group 3 volunteers received Dimolegin (DD217) once at a dose of 60 mg
  Interventions: Drug: Dimolegin

INTERVENTIONS:
Drug: Dimolegin — Dimolegin (DD217) - enteric coated tablets 10 mg developed by PharmaDiall Ltd (Moscow), manufactured by Federal State Unitary Enterprise Research and Practical Center "Pharmaceutical Protection" at The Federal Medical Biological Agency (FMBA) of Russia
  Other Names: DD217

SUMMARY:
In the course of the clinical study, the pharmacokinetics, pharmacodynamics, safety and tolerability of Dimolegin (DD217) 10 mg enteric-coated tablets after single administration to healthy volunteers at increasing doses were studied.

24 volunteers participated in the study. The randomization procedure was carried out for 24 volunteers selected at screening. In Group 1 6 volunteers were randomized , in Group 2 6 volunteers were randomized, and in Group 3 12 volunteers were enrolled. Group 1 volunteers took the study drug at a dose of 20 mg once, group 2 volunteers took the study drug at a dose of 40 mg once, and group 3 volunteers took the study drug at a dose of 60 mg once.

DETAILED DESCRIPTION:
Study objectives were:

1. to evaluate the safety of different single doses of Dimolegin (DD217) in healthy volunteers;
2. to evaluate the tolerance of different single doses of Dimolegin (DD217) in healthy volunteers;
3. to evaluate pharmacokinetic parameters with a single dose of Dimolegin (DD217) in increasing doses;
4. to evaluate the effect of Dimolegin (DD217) on coagulation profile parameters (prothrombin time, activated partial thromboplastin time (aPTT), anti-Xa activity) with a single dose in healthy volunteers (pharmacodynamic study).

Study design was an open study of the pharmacokinetics, safety and tolerability of Dimolegin (DD217) after single administration to healthy volunteers in fasting conditions (phase 1).

Study population was: screened - 40, randomized - 24, per protocol population - 24.

The study was open, prospective, non-randomized with sequential enrollment of volunteers with dose escalation Group No. 1 (n=6) consisted of 2 cohorts with 3 volunteers per each. Volunteers of Cohorts 1 and 2 received Dimolegin (DD217) once at a dose of 20 mg.

Group No. 2 (n=6) consisted of 2 cohorts with 3 volunteers per each. Volunteers of Cohorts 3 and 4 received Dimolegin (DD217) once at a dose of 40 mg.

Group No. 3 (n=12) consisted of 3 cohorts. Cohorts 5 and 6 included 3 volunteers per each, and Cohort 7 included 6 volunteers. All Group 3 volunteers received Dimolegin (DD217) once at a dose of 60 mg.

Initially, the first cohort (n=3) of volunteers was included in the study, in which volunteers received the study drug once at a dose of 20 mg. After evaluation of the interim safety results (complete blood count and blood chemistry, urinalysis, clinical health assessment, electrocardiogram (ECG)) 3 days after dosing in the absence of SAEs, the Investigator decided to include the second cohort (n=3), in which volunteers continued to receive the drug at a single dose of 20 mg.

28 days after dosing in Cohort 2 of Group 1, the Investigator compiled a report on the safety of the study drug dose based on the results of all safety tests (complete blood count and blood chemistry, urinalysis), ECG and clinical health assessment, based on the submitted IDMC report, a decision was made to enroll volunteers to Group 2, also consisting of 2 cohorts: the third and the fourth.

Volunteers of Group 2, Cohort 3 (n=3) received a single study drug dose of 40 mg. After evaluation of the interim safety results (complete blood count and blood chemistry, urinalysis, clinical health assessment, ECG) 3 days after dosing in the absence of SAEs, the Investigator decided to include the forth cohort (n=3), in which volunteers continued to take the drug at a single dose of 40 mg. 28 days after dosing in Cohort 4 of Group 2, the Investigator compiled a report on the safety of the study drug dose based on the results of all safety tests (complete blood count and blood chemistry, urinalysis), ECG and clinical health assessment, based on the submitted IDMC report, a decision was made to enroll volunteers to Group 3, also consisting of 3 cohorts: the fifth, the sixth and the seventh.

The volunteers of Group 3, Cohort 5 (n=3), took a single study drug dose of 60 mg. After evaluation of the interim safety results (complete blood count and blood chemistry, urinalysis, clinical health assessment, ECG) 3 days after dosing in the absence of SAEs, the Investigator decided to include the sixth cohort (n=3), in which volunteers continued to take the drug at a single dose of 60 mg. 28 days after dosing in Cohort 6 of Group 3, the Investigator compiled a report on the safety of the study drug dose based on the results of all safety tests (complete blood count and blood chemistry, urinalysis), ECG and clinical health assessment, based on the submitted IDMC report, a decision was made to enroll volunteers to Cohort 7 (n=6) of Group 3. Cohort 7 volunteers continued to take 60 mg of the study drug orally once and completed the study.

In chronic toxicity studies, adverse effects were achieved on Day 42 in rats at a dose of 90 mg/kg of DD217 substance and on Day 46 in rabbits at a dose of 100 mg/kg of DD217 substance, which, after conversion to maximum recommended starting dose (MRSD) for human, gave 0.60 mg/kg and 1.56 mg/kg, respectively. These doses were considered as an estimate of the upper limit of dose, that is, the MRSD should have been less than 0.60 mg/kg. Thus, 0.28 mg/kg was taken as MRSD, i.e. in terms of a person weighing 70 kg, MRSD = 0.28*70 = 20 mg as a single dose. To ensure the safety of volunteers, the study was performed with a phased dose escalation. Given Cmax and T1/2 values, in the absence of any SAEs, dosing in the next cohort should be no earlier than 3 days after the drug is given to the previous cohort. In the case of SAE dosing in the next cohort could be performed only after approval by an Independent Data Monitoring Committee (IDMC - created before the start of the study, the composition of 3 experts is approved by the Local Ethics Committee). Dose escalation (switch to the next group) was possible no earlier than 28 days after the last dosing in the study group and with the approval of the IDMC.

The study drug was used once in the morning in fasting state. Clinical assessment of health state (physical examination and measurement of vital signs (blood pressure, heart rate, respiratory rate, body temperature), laboratory parameters (complete blood count, blood cell morphology differentials, blood chemistry, urinalysis) were determined in accordance with the set goal and objectives.

Blood coagulation profile parameters (prothrombin time, APTT and anti-Xa activity) were determined for construction of pharmacodynamic curves in discrete time intervals in accordance with the set goal and objectives.

Dioxaban (DD217) concentration was determined in discrete time intervals in accordance with the set goal for the construction of pharmacokinetic curves based on which, in turn, the pharmacokinetic parameters of the active substances were calculated.

Pharmacokinetic parameters were calculated by a model-independent method. The following parameters were calculated for all the subjects:

AUCo-t- area under concentration-time curve from 0 to the last blood sampling; AUCo-inf-area under concentration-time curve (from 0 to infinity); Cmax- maximum concentration value; Tmax- time to maximum concentration; T1/2-half-life; Cl - clearance. Study duration Maximum duration for each volunteer did not exceed 42 days. Descriptive statistics was provided for all demographic and other baseline characteristics, safety parameters and their changes (if applicable) in course of the study by time points of evaluation and by groups. Descriptive statistics for quantitative variables included mean, median, standard deviation, minimum and maximum values, and the number of observations. Qualitative data are presented as frequencies and proportions in percentage terms. The baseline values for laboratory, instrumental and vital safety parameters were the values obtained at Visit 0 (Screening) or at Visit 1 before dosing.

Per Protocol (PP) population included all volunteers for the assessment of pharmacodynamics and pharmacokinetics who met the inclusion/exclusion criteria and received the prescribed dose of the study drug. There were no volunteers who withdrew from this study.

When planning the sample size for an experimental study, the number of 24 healthy volunteers was recognized as acceptable. Due to the descriptive nature of this study, the sample size determination was not based on any formal statistical assumptions.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-45 years
* Verified "healthy" diagnosis based on the findings of routine clinical, laboratory, and instrumental examinations
* Body mass index (BMI) is 18.5-30.0 kg/m2
* Consent to the use of barrier contraception methods during the study period and for 3 months after it
* Written consent of the volunteer to enrollment

Exclusion Criteria:

* Aggravated allergy history
* Drug intolerance
* Acute and chronic cardiovascular, bronchopulmonary, neuroendocrine diseases as well as gastrointestinal, hepatic, renal, hematological diseases
* Systolic blood pressure less than 90 mmHg or above 130 mmHg
* Diastolic blood pressure less than 70 mmHg or above 89 mmHg
* Pulse rate less than 60 bpm or more than 89 bpm
* Gastrointestinal surgery (except for appendectomy)
* Acute infectious diseases less than 4 weeks prior to the study
* Any abnormalities detected during screening from the clinical laboratory center reference values (including estimated glomerular filtration rate (GFR), coagulation profile), clinical and instrumental study methods
* Hypersensitivity to the study product components
* Taking prescription or over-the-counter medications, including dietary supplements, herbal products, vitamins, homeopathic medicines, less than 2 weeks before the start of the study
* Administration of medicinal products with expressed effect on hemodynamics, hepatic function and other systems (e.g. barbiturates, omeprazole, cimetidine, etc.) less than 2 months prior to the study initiation
* Blood donation (≥ 450 mL of blood or plasma) less than 2 months prior to the study
* Participation in clinical studies of drug products less than 3 weeks prior to the study initiation
* Intake of more than 10 units of alcohol per week (10 mL of pure (100 %) ethanol is taken for 1 unit of alcohol, this is the amount that the body of a healthy adult breaks down within an hour; 1 unit of alcohol is equivalent to 0.33 liters of beer, 150 mL of wine or 30 mL of hard liquors), or history of alcohol or drug dependence, drug abuse
* Smoking > 10 cigarettes per day
* Positive urine drug test (cocaine, cannabis, amphetamines, barbiturates and opioids)
* Positive alcohol breath test
* Lost for follow-up during 29 days, inability to comply with the schedule of visits, inability to be hospitalized for 2.5 days
* Inability to understand or follow protocol instructions

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 24 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2017-12-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Total Adverse Events (AE) | 28 Days
  Number of of subjects experiencing AEs, serious adverse events (SAEs), or discontinuations due to AEs

SECONDARY OUTCOMES:
The increase in Anti-Xa activity | 2 Days
  The maximum increase in Anti-Xa activity after Dimolegin administration. Anti-Xa values are averaged over all subjects in the group.
The increase in International Normalised Ratio (INR) | 2 Days
  The maximum increase in INR after Dimolegin administration. INR values are averaged over all subjects in the group.
The increase in Activated Partial Thromboplastin Time (aPTT) | 2 Days
  The maximum increase in aPTT after Dimolegin administration. aPTT values are averaged over all subjects in the group.
Steady-state Area Under the Plasma Concentration Versus Time Curve From Time Zero to 12 Hours of Dioxaban (AUC (0-12)) | 7 Days
  Area Under the Curve AUC (0-12) is the area under the curve from time 0 to 12 hour after dioxaban steady state concentration is reached.
Steady state Elimination of Half-Life of Dioxaban (t½) | 7 Days
  Mean terminal phase plasma t½ of dioxaban at steady-state
Steady-state Maximum Observed Plasma Concentration of Dioxaban (Cmax) | 7 Days
  Maximum observed drug concentration in plasma after administration Cmax of dioxaban at steady-state
Steady state Plasma Clearance of Dioxaban (CL) | 7 Days
  CL of dioxaban at steady-state
Steady-state Time to Maximum Observed Plasma Concentration of Dioxaban | 7 Days
  Time to Maximum observed drug concentration in plasma after administration (Tmax) of dioxaban at steady-state

CONTACTS AND LOCATIONS:
Locations (1):
- Non-Governmental Private Healthcare Institution of Sci-entific Clinical Center of Russian Railways JSC, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tovbin DG, Tarasov DN, Malakhov DV, Tserkovnikova NA, Aybush AV, Drozd NN. The Development of New Low-Molecular-Weight Factor Xa Inhibitors that are Potential Anticoagulants. Curr Drug Discov Technol. 2022;19(1):e010921191770. doi: 10.2174/1568009621666210224104940. PMID 33655836
- [Background] Tarasov DN, Tovbin DG, Malakhov DV, Aybush AV, Tserkovnikova NA, Savelyeva MI, Sychev DA, Drozd NN, Savchenko AY. The Development of New Factor Xa Inhibitors Based on Amide Synthesis. Curr Drug Discov Technol. 2018;15(4):335-350. doi: 10.2174/1570163815666180215114732. PMID 29468977